CLINICAL TRIAL: NCT03523247
Title: A Whole Food, Plant Based Diet and Its Lipidemic Effects on Primary Prevention Population in a Free-range Environment - a Pilot Study
Brief Title: A Whole Food Plant Diet and Its Lipidemic Effects on Primary Prevention in a Free-range Population
Acronym: WholeLIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lancaster General Hospital (Other)
Collaborators: Louise von Hess Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYP2018_CW0001
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Diet Modification; Cardiology
Keywords: Cholesterol; LDL; HDL; triglycerides; c-reactive protein; whole food diet; plant based diet; community based enrollment
MeSH Terms: interventions — Diet, Plant-Based

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole Food Plant Based Diet (Experimental): Single-arm whole-food, plant-based diet will explore the effects on primary prevention in a free-range environment
  Interventions: Behavioral: whole food, plant based diet

INTERVENTIONS:
Behavioral: whole food, plant based diet — whole food, plant based diet featuring vegetables, fruits, legumes, whole grains, seeds, and nuts

SUMMARY:
This study seeks to determine the effects of a whole-food, plant-based diet on lipid, metabolic, and inflammatory biomarkers. Eligible participants will have had either an LDL-C >100 mg/dL or non-HDL-C >130 mg/dL without a current diagnosis of coronary heart disease and are willing to adhere to a whole food plant based diet for at least 8 weeks. Participants enrolled in the study will provide fasting blood work, complete a baseline quality of life survey, and receive education on a whole-food, plant-based diet at a local Lancaster County grocery store during their first study visit. Throughout the study, patients will have access to dietary counseling which will be provided by a certified nutritionist and will be asked to record and submit daily food diaries. Study participants will be asked to adhere to a whole food plant based diet for a total of 8 weeks. Prior to the final study visit, participants will be asked to obtain follow-up fasting bloodwork around 7 weeks post start of whole food plant based diet. The results, along with a follow-up quality of life survey, and an opportunity to discuss the bloodwork with a doctor will be held at the local grocery story 8 weeks after the first study visit.

DETAILED DESCRIPTION:
CHD remains the leading cause of death in numerous developed countries and is estimated to cause one-third of all deaths in patients over the age of 35. 28 While CVD is preventable, studies suggest that a range of lifestyle factors including physical inactivity, nicotine abuse, and nutrition practices are increasing the prevalence of the disease in most countries. 28,29 Such facts highlight the importance of lifestyle interventions. Despite the chronic nature of cardiovascular disease, even short-term studies analyzing ad libitum plant-based diets reveal significantly improved changes in commonly tested biomarkers that predict cardiovascular disease risk. 30 While a number of studies have explored the lipid-lowering effects of traditional vegetarian diets, 31 few studies have explored the effects of a whole-food, plant-based diet despite its proposed benefits. Preliminary studies suggest that such a diet might facilitate weight loss and lead to improvements in lipid parameters.32 To this end, we propose a study to implement a whole-food, plant based diet intervention in the Lancaster community to quantify its ability to modify lipid, metabolic and inflammatory biomarkers.

This single-arm diet pilot study seeks to determine the serologic effects of a whole-food, plant-based diet on primary prevention subjects in a free-range environment. Eligible participants will have had either an LDL-C >100 mg/dL or non-HDL-C >130 mg/dLwithout a current diagnosis of coronary heart disease and are willing to adhere to a whole food plant based diet for at least 8 weeks.

A total of 50 subjects will be enrolled to the study. Participants enrolled in the study will provide fasting blood work and receive education on a whole-food, plant-based diet at a local Lancaster County grocery store during their first study visit. At this time, the study coordinator will also document the patient's height, weight, and hip and waist circumference. While subjects are waiting to provide a blood draw, study personnel will administer two baseline questionnaires to each subject. The first questionnaire will be the SF12 quality-of-life survey. The second survey will capture pertinent elements of the patient's medical history and ask the patient questions on motivation, attitude, and expected compliance to the diet.They will be served a catered vegan breakfast and receive a lecture on a whole-food, plant-based diet by Dr. Christopher Wenger. Dr. Wenger also will train the subjects on the use of the study food record. At the end of the session, a certified nutritionist will give a tour of the local grocery store to show subjects how to select appropriate low-cost foods for the dietary intervention. Following the conclusion of the study visit, subjects will begin the interventional phase of the study and follow a whole-food, plant-based diet for eight weeks. The dietary intervention will conclude with the post-intervention study visit. Throughout the study, patients will have access to dietary counseling which will be provided by a certified nutritionist

The post-intervention study visit (8 weeks after the initial visit) will be held at the conference room in the local grocery story and will comprise the same cohort which began the study together at the baseline study visit. Prior to distributing each subject's results, study personnel will administer the SF12 quality-of-life survey and measure each subject's weight and hip and waist circumference post-intervention. Study personnel will also administer a questionnaire assessing each subject's experience on the diet including challenges, motivation, and attitudes toward the diet. We will also capture how likely the patient is to continue on the diet after the conclusion of the study.

Study personnel will then disseminate each patient's lab results pre- and post-intervention. At this time, subjects will be given the opportunity to discuss their results with Dr. Wenger. A catered vegan lunch will be served during the study visit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Indicated willingness to adhere to whole-food plant-based diet
* Patient recommended for dietary intervention by healthcare provider
* LDL-C >100 mg/dL or non-HDL-C >130 mg/dL documented by a lab test in the LG EMR within the last 6 months

Exclusion Criteria:

* Any condition that, in the opinion of the patient's healthcare provider, will adversely affect study execution or data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Percent change in cholesterol specific biomarkers | from baseline (study one visit) through 7 weeks of diet change
  Percent change in LDL cholesterol, non-HDL cholesterol, and LDL particle concentration from baseline values

SECONDARY OUTCOMES:
Percent change in cholesterol specific biomarkers | from baseline (study one visit) through 7 weeks of diet change
  Percent change in triglyceride concentration
Percent change in specific cholesterol biomarkers | from baseline (study one visit) through 7 weeks of diet change
  Percent change in lipoprotein(a)
Percent change in inflammatory biomarkers | from baseline (study one visit) through 7 weeks of diet change
  Percent change in C-reactive protein
Dietary behavioral modifications and adherence | from baseline (study one visit) through 7 weeks of diet change
  Evaluation of changes made to diet and their respective adherence over time

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Wenger, DO, Principal Investigator — Penn Medicine/Lancaster General Health
Locations (1):
- Penn Medicine / Lancaster General Hospital, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] US Department of Health and Human Services. The surgeon general's call to action to prevent and decrease overweight and obesity. Rockville, MD: US Department of Health and Human Services, Public Health Service, Office of the Surgeon General; 2001 [cited 22 Jan 2013].
- [Background] Reedy J, Krebs-Smith SM, Miller PE, Liese AD, Kahle LL, Park Y, Subar AF. Higher diet quality is associated with decreased risk of all-cause, cardiovascular disease, and cancer mortality among older adults. J Nutr. 2014 Jun;144(6):881-9. doi: 10.3945/jn.113.189407. Epub 2014 Feb 26. PMID 24572039
- [Background] McCullough ML. Diet patterns and mortality: common threads and consistent results. J Nutr. 2014 Jun;144(6):795-6. doi: 10.3945/jn.114.192872. Epub 2014 Apr 9. No abstract available. PMID 24717365
- [Background] Berkow SE, Barnard N. Vegetarian diets and weight status. Nutr Rev. 2006 Apr;64(4):175-88. doi: 10.1111/j.1753-4887.2006.tb00200.x. PMID 16673753
- [Background] Farmer B, Larson BT, Fulgoni VL 3rd, Rainville AJ, Liepa GU. A vegetarian dietary pattern as a nutrient-dense approach to weight management: an analysis of the national health and nutrition examination survey 1999-2004. J Am Diet Assoc. 2011 Jun;111(6):819-27. doi: 10.1016/j.jada.2011.03.012. PMID 21616194